CLINICAL TRIAL: NCT05370300
Title: Subtraction Normalized Aggregated Phagocytic Signal in Peripheral Blood of Breast Cancer Patients (SNAPS - Clinical Trial) A NextGen RNASeq Feasibility Study of a Blood-based Model for Early Cancer Detection and Surveillance
Brief Title: SNAPS Breast Cancer Patient Study Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Immunis.AI (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: SNAPS Breast Cancer
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: Breast Cancer; Immunogenomics
MeSH Terms: conditions — Breast Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Patients with negative screening MMG: Patients presenting to Duke Radiology for routine screening mammogram will be screened for eligibility as negative controls. Study enrollment for negative controls presumes that patients do not receive their screening mammography results immediately. Patients will be approached on the day of their first new patient visit to the Duke Cancer Center. If they are willing, they will be consented in clinic, and directed down to the lab for their first blood draw.
  Interventions: Diagnostic Test: Blood test
- Cases: Patients with known cancer diagnosis: Patients presenting to the Duke Cancer Center for evaluation by Medical or Surgical Oncology of a newly diagnosed breast cancer will be screened for study eligibility and approached, enrolled, and consented accordingly. Patients will be approached on the day of their first new patient visit to the Duke Cancer Center. If they are willing, they will be consented in clinic, and directed down to the lab for their first blood draw.
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Proprietary immunogenomic signature from peripheral blood CD14 and CD2 cells.

SUMMARY:
Differential immunogenomic signatures from peripheral blood CD14 (phagocytic) and CD2 (non-phagocytic) cells have been associated with multiple cancers and disease states. In particular several large clinical studies at Immunis.AI have demonstrated robust immunogenomic signatures in early-stage prostate cancer. Immunis.AI therefore hypothesizes that a peripheral blood immunogenomic signature will identify patients with various stages of breast cancer from healthy negative controls.

DETAILED DESCRIPTION:
Efficient next generation RNA sequencing platforms have allowed for whole genome expression profiling of individual populations of immune cells as a novel means of searching for patterns of gene expression to aid in the identification of meaningful signals unique to various disease states. Single cell sequencing techniques have provided additional information useful in deconvolution strategies applied to model development on purified populations of immune cells. Recent interest in peripheral leukocyte subset gene expression profiles suggests that diagnostic information for many disorders may be contained therein. Mononuclear phagocytic cells including the various CD14+ subsets have been studied extensively in various disease states including some solid tumors. Previous large clinical studies at Immunis.AI have determined that transcriptomic profiles of CD14+ cell populations subtraction normalized from CD2+ cell populations were associated with aggressive disease phenotypes such as prostate cancer. Tumor heterogeneity, multifocality, and oligoclonality have been a significant barrier to development of meaningful tissue based multigene signatures for predicting cancer biologic behavior. The findings at Immunis.AI strongly suggest that analysis of RNA expression data from the body's immune surveillance cells has the potential to summarize the entire heterogeneous tumor. The investigators believe that the CD14/CD2 log ratio can be understood as a subtraction normalization of gene expression which yields superior signal of early-stage cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 yrs of age.
* Patients diagnosed with stage I-IV breast cancer, who have not begun definitive therapy.
* Patients undergoing screening mammograms for breast cancer.

Exclusion Criteria:

* Patients with a history of a different cancer within the previous 3 years (except non melanoma skin cancer).
* Any prior treatment (surgery, chemo, hormonal, radiation, biologics, etc.) for current cancer.
* Any biopsy which resulted in the entire tumor tissue being removed.
* History of previous breast cancer.
* Patients unable to provide informed consent.
* Patients with an abnormal screening mammogram.
* Patients whose hormone receptor and/or HER2 status are not available.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Duke Cancer Center for evaluation by Medical or Surgical Oncology of a newly diagnosed breast cancer Patients presenting to Duke Radiology for routine screening mammogram
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Aim | 12 months
  To determine if differential gene expression between peripheral blood phagocytic and non-phagocytic immune cells can distinguish breast cancer patients from cancer-negative controls.

SECONDARY OUTCOMES:
Secondary Aim 1 | 12 months
  To evaluate minimal residual disease with a potential signature for breast cancer detection following curative therapy to evaluate the degree to which the original signature has changed.
Secondary Aim 2 | 12 months
  To determine the sample size required to develop and validate a computational immunogenomic model capable of predicting the various types, grades, and stages of breast cancer.
Secondary Aim 3 | 12 months
  To determine the temporal relation between biopsy procedures and signal strength or dilution.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Wojno, MD, Principal Investigator — Immunis.AI
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Research data will not be shared as it is proprietary information

REFERENCES:
- [Result] Van Neste L, Wojno KJ, Henao R, Mane S, Korman H, Hafron J, Kernen K, Tinawi-Aljundi R, Putzi M, Kassis AI, Kantoff PW. Evaluation of an RNAseq-Based Immunogenomic Liquid Biopsy Approach in Early-Stage Prostate Cancer. Cells. 2021 Sep 28;10(10):2567. doi: 10.3390/cells10102567. PMID 34685549
- [Result] Palmer C, Diehn M, Alizadeh AA, Brown PO. Cell-type specific gene expression profiles of leukocytes in human peripheral blood. BMC Genomics. 2006 May 16;7:115. doi: 10.1186/1471-2164-7-115. PMID 16704732
- [Result] Schmidl C, Renner K, Peter K, Eder R, Lassmann T, Balwierz PJ, Itoh M, Nagao-Sato S, Kawaji H, Carninci P, Suzuki H, Hayashizaki Y, Andreesen R, Hume DA, Hoffmann P, Forrest AR, Kreutz MP, Edinger M, Rehli M; FANTOM consortium. Transcription and enhancer profiling in human monocyte subsets. Blood. 2014 Apr 24;123(17):e90-9. doi: 10.1182/blood-2013-02-484188. Epub 2014 Mar 26. PMID 24671955
- [Result] Hashimoto S, Nagai S, Sese J, Suzuki T, Obata A, Sato T, Toyoda N, Dong HY, Kurachi M, Nagahata T, Shizuno K, Morishita S, Matsushima K. Gene expression profile in human leukocytes. Blood. 2003 May 1;101(9):3509-13. doi: 10.1182/blood-2002-06-1866. Epub 2003 Jan 9. PMID 12522010
- [Result] Dale DC, Boxer L, Liles WC. The phagocytes: neutrophils and monocytes. Blood. 2008 Aug 15;112(4):935-45. doi: 10.1182/blood-2007-12-077917. PMID 18684880
- [Result] Gutknecht MF, Bouton AH. Functional significance of mononuclear phagocyte populations generated through adult hematopoiesis. J Leukoc Biol. 2014 Dec;96(6):969-80. doi: 10.1189/jlb.1RI0414-195R. Epub 2014 Sep 15. PMID 25225678
- [Result] Chow A, Brown BD, Merad M. Studying the mononuclear phagocyte system in the molecular age. Nat Rev Immunol. 2011 Oct 25;11(11):788-98. doi: 10.1038/nri3087. PMID 22025056
- [Result] Epstein JI. Update on the Gleason grading system. Ann Pathol. 2011 Nov;31(5 Suppl):S20-6. doi: 10.1016/j.annpat.2011.08.023. Epub 2011 Sep 28. No abstract available. PMID 22054451
- [Result] Grignon DJ. Prostate cancer reporting and staging: needle biopsy and radical prostatectomy specimens. Mod Pathol. 2018 Jan;31(S1):S96-109. doi: 10.1038/modpathol.2017.167. PMID 29297497
- [Result] Boutros PC, Fraser M, Harding NJ, de Borja R, Trudel D, Lalonde E, Meng A, Hennings-Yeomans PH, McPherson A, Sabelnykova VY, Zia A, Fox NS, Livingstone J, Shiah YJ, Wang J, Beck TA, Have CL, Chong T, Sam M, Johns J, Timms L, Buchner N, Wong A, Watson JD, Simmons TT, P'ng C, Zafarana G, Nguyen F, Luo X, Chu KC, Prokopec SD, Sykes J, Dal Pra A, Berlin A, Brown A, Chan-Seng-Yue MA, Yousif F, Denroche RE, Chong LC, Chen GM, Jung E, Fung C, Starmans MH, Chen H, Govind SK, Hawley J, D'Costa A, Pintilie M, Waggott D, Hach F, Lambin P, Muthuswamy LB, Cooper C, Eeles R, Neal D, Tetu B, Sahinalp C, Stein LD, Fleshner N, Shah SP, Collins CC, Hudson TJ, McPherson JD, van der Kwast T, Bristow RG. Spatial genomic heterogeneity within localized, multifocal prostate cancer. Nat Genet. 2015 Jul;47(7):736-45. doi: 10.1038/ng.3315. Epub 2015 May 25. PMID 26005866
- [Result] Womble PR, Montie JE, Ye Z, Linsell SM, Lane BR, Miller DC; Michigan Urological Surgery Improvement Collaborative. Contemporary use of initial active surveillance among men in Michigan with low-risk prostate cancer. Eur Urol. 2015 Jan;67(1):44-50. doi: 10.1016/j.eururo.2014.08.024. Epub 2014 Aug 24. PMID 25159890
- [Result] Cher ML, Dhir A, Auffenberg GB, Linsell S, Gao Y, Rosenberg B, Jafri SM, Klotz L, Miller DC, Ghani KR, Bernstein SJ, Montie JE, Lane BR; Michigan Urological Surgery Improvement Collaborative. Appropriateness Criteria for Active Surveillance of Prostate Cancer. J Urol. 2017 Jan;197(1):67-74. doi: 10.1016/j.juro.2016.07.005. Epub 2016 Jul 14. PMID 27422298